CLINICAL TRIAL: NCT01707992
Title: A Multinational, Multicenter, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled Study Followed by an Active Treatment Period, to Evaluate the Efficacy, Safety and Tolerability of Two Doses of Oral Administration of Laquinimod (0.6 mg/Day or 1.2 mg/Day) in Patients With Relapsing Remitting Multiple Sclerosis (RRMS)
Brief Title: The Efficacy, Safety, and Tolerability of Laquinimod in Participants With Relapsing Remitting Multiple Sclerosis (RRMS)
Acronym: CONCERTO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LAQ-MS-305; 2012-003647-30 (EudraCT Number)
Record Dates: First submitted 2012-09-28; First posted 2012-10-16 (Estimated); Results first posted 2019-03-13 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — laquinimod

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Placebo-Controlled Phase: Placebo (Placebo Comparator): Participants will receive 2 capsules of placebo (matching to laquinimod 0.6 milligrams [mg]) once daily orally for up to 24 months.
  Interventions: Drug: Placebo
- Placebo-Controlled Phase: Laquinimod 0.6 mg (Experimental): Participants will receive 1 capsule of laquinimod 0.6 mg and 1 capsule of matching placebo once daily orally for up to 24 months.
  Interventions: Drug: Laquinimod; Drug: Placebo
- Placebo-Controlled Phase: Laquinimod 1.2 mg (Experimental): Participants will receive laquinimod 1.2 mg (2 capsules of laquinimod 0.6 mg each) once daily orally for up to 24 months.
  Interventions: Drug: Laquinimod
- Active Treatment Phase: Laquinimod 0.6 mg (Experimental): Participants who completed the placebo-controlled phase on placebo and on laquinimod 0.6 mg treatment group after 01 January 2016, will receive 1 capsule of laquinimod 0.6 mg and 1 capsule of matching placebo once daily orally for 24 months.
  Interventions: Drug: Laquinimod; Drug: Placebo
- Active Treatment Phase: Laquinimod 1.2 mg (Experimental): Participants who completed the placebo-controlled phase on placebo and on laquinimod 1.2 mg treatment group prior to 01 January 2016, will receive laquinimod 1.2 mg (2 capsules of laquinimod 0.6 mg each) once daily orally for 24 months.
  Interventions: Drug: Laquinimod
- Active Treatment Phase: Off Drug (No Intervention): Participants who were discontinued from treatment with laquinimod 1.2 mg during the placebo-controlled phase due to sponsor decision after 01 January 2016 will continue the active-treatment phase off drug for 24 months.

INTERVENTIONS:
Drug: Laquinimod — Laquinimod will be administered as per the dose and schedule specified in the respective arms.
  Arms: Active Treatment Phase: Laquinimod 0.6 mg; Active Treatment Phase: Laquinimod 1.2 mg; Placebo-Controlled Phase: Laquinimod 0.6 mg; Placebo-Controlled Phase: Laquinimod 1.2 mg
Drug: Placebo — Placebo matching to laquinimod will be administered as per the schedule specified in the respective arms.
  Arms: Active Treatment Phase: Laquinimod 0.6 mg; Placebo-Controlled Phase: Laquinimod 0.6 mg; Placebo-Controlled Phase: Placebo

SUMMARY:
This is a multinational, multicenter, randomized, double-blind, parallel-group, placebo-controlled study followed by active treatment, to evaluate the efficacy, safety and tolerability of two doses of oral administration of laquinimod in participants with RRMS. The study has 2 periods: Period 1, the double-blind, placebo-controlled period (up to 24 months) and Period 2, the active treatment period (24 months).

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a confirmed and documented multiple sclerosis (MS) diagnosis as defined by the Revised McDonald criteria, with relapse onset disease or a relapsing-remitting disease course.
* Participants must be ambulatory with Kurtzke's expanded disability status scale (EDSS) score of 0 to 5.5 in both screening and randomization visits.
* Participants must be in a stable neurological condition, relapse-free and free of any corticosteroid treatment [intravenous (IV), intramuscular (IM) and/or per os (PO)/oral] or adrenocorticotrophic hormone, 60 days prior to randomization.
* Participants must have experienced at least one documented relapse in the 12 months prior to randomization.
* Participants must have disease duration of not more than 15 years.
* Women of child-bearing potential (for example, women who are not postmenopausal or surgically sterilized) must practice an acceptable method of birth control for 30 days before taking the study drug and two acceptable methods of birth control during the duration of the study and until 30 days after the last dose of study medication.

  * Additional criteria apply, please contact the investigator for more information.

Exclusion Criteria:

* Participants with progressive forms of MS.
* Participants with neuromyelitis optica.
* Use of experimental or investigational drugs and/or participation in drug clinical studies within the 6 months prior to randomization.
* Use of immunosuppressive agents or cytotoxic agents, including cyclophosphamide, within 6 months prior to randomization.
* Use of either of the following within 2 years prior to randomization visit: natalizumab (Tysabri®), rituximab, ocrelizumab, atacicept, belimumab, or ofatumumab.
* Use of teriflunomide (Aubagio®) within 2 years prior to randomization, except if active washout (with either cholestyramine or activated charcoal) was done 2 months or more prior to randomization.
* Previous treatment with glatiramer acetate (Copaxone®) Interferon β (either 1a or 1b), fingolimod (Gilenya®), dimethyl fumarate (Tecfidera®) or intravenous immunoglobulins within 2 months prior to randomization.
* Chronic (more than 30 consecutive days) systemic (IV, IM or PO) corticosteroid treatment within 2 months prior to randomization.
* Previous use of mitoxantrone (Novantrone®), cladribine, or alemtuzumab (Lemtrada®).
* Previous use of laquinimod.
* Previous total body irradiation or total lymphoid irradiation.
* Previous stem cell treatment, autologous bone marrow transplantation or allogenic bone marrow transplantation.
* Use of moderate/strong inhibitors of cytochrome P450 (CYP) 3A4 within 2 weeks prior to randomization.
* Use of inducers of CYP3A4 within 2 weeks prior to randomization visit.
* Pregnancy or breastfeeding.
* A known history of sensitivity to gadolinium (Gd).
* Inability to successfully undergo magnetic resonance imaging (MRI) scanning.
* Participants who underwent endovascular treatment for chronic cerebrospinal venous insufficiency within 3 months prior to randomization.

  * Additional criteria apply, please contact the investigator for more information.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2199 (Actual)
Dates: Start 2013-02-20 (Actual); Primary Completion 2015-04-13 (Actual); Study Completion 2017-07-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (284):
- United States (32):
  - Teva Investigational Site 10329, Cullman, Alabama
  - Teva Investigational Site 10349, Sun City, Arizona
  - Teva Investigational Site 10342, Tucson, Arizona
  - Teva Investigational Site 10310, Fresno, California
  - Teva Investigational Site 10307, Aurora, Colorado
  - Teva Investigational Site 10334, Centennial, Colorado
  - Teva Investigational Site 10332, Fort Collins, Colorado
  - Teva Investigational Site 10316, Coral Gables, Florida
  - Teva Investigational Site 10308, Sarasota, Florida
  - Teva Investigational Site 10341, St. Petersburg, Florida
  - Teva Investigational Site 10315, Sunrise, Florida
  - Teva Investigational Site 10323, Tampa, Florida
  - Teva Investigational Site 10350, Chicago, Illinois
  - Teva Investigational Site 10345, Evanston, Illinois
  - Teva Investigational Site 10343, Northbrook, Illinois
  - Teva Investigational Site 10339, Fort Wayne, Indiana
  - Teva Investigational Site 10348, Lenexa, Kansas
  - Teva Investigational Site 10338, Boston, Massachusetts
  - Teva Investigational Site 10346, Advance, North Carolina
  - Teva Investigational Site 10347, Winston-Salem, North Carolina
  - Teva Investigational Site 10309, Bellevue, Ohio
  - Teva Investigational Site 10317, Columbus, Ohio
  - Teva Investigational Site 10325, Dayton, Ohio
  - Teva Investigational Site 10340, Hershey, Pennsylvania
  - Teva Investigational Site 10331, Philadelphia, Pennsylvania
  - Teva Investigational Site 10313, Cordova, Tennessee
  - Teva Investigational Site 10324, Franklin, Tennessee
  - Teva Investigational Site 10318, Nashville, Tennessee
  - Teva Investigational Site 10319, Salt Lake City, Utah
  - Teva Investigational Site 10330, Newport News, Virginia
  - Teva Investigational Site 10311, Roanoke, Virginia
  - Teva Investigational Site 10335, Seattle, Washington
- Austria (4):
  - Teva Investigational Site 33013, Innsbruck
  - Teva Investigational Site 33014, Linz
  - Teva Investigational Site 33016, Vienna
  - Teva Investigational Site 33015, Vienna
- Belarus (6):
  - Teva Investigational Site 68013, Grodno
  - Teva Investigational Site 68010, Homyel
  - Teva Investigational Site 68012, Minsk
  - Teva Investigational Site 68009, Minsk
  - Teva Investigational Site 68008, Minsk
  - Teva Investigational Site 68011, Vitebsk
- Belgium (2):
  - Teva Investigational Site 37023, Charleroi
  - Teva Investigational Site 37024, Sijsele
- Bosnia and Herzegovina (3):
  - Teva Investigational Site 69008, Mostar
  - Teva Investigational Site 69006, Sarajevo
  - Teva Investigational Site 69009, Tuzla
- Bulgaria (24):
  - Teva Investigational Site 59039, Pleven
  - Teva Investigational Site 59040, Pleven
  - Teva Investigational Site 59060, Pleven
  - Teva Investigational Site 59062, Plovdiv
  - Teva Investigational Site 59061, Rousse
  - Teva Investigational Site 59055, Shumen
  - Teva Investigational Site 59048, Sofia
  - Teva Investigational Site 59052, Sofia
  - Teva Investigational Site 59057, Sofia
  - Teva Investigational Site 59050, Sofia
  - Teva Investigational Site 59044, Sofia
  - Teva Investigational Site 59063, Sofia
  - Teva Investigational Site 59038, Sofia
  - Teva Investigational Site 59043, Sofia
  - Teva Investigational Site 59058, Sofia
  - Teva Investigational Site 59041, Sofia
  - Teva Investigational Site 59042, Sofia
  - Teva Investigational Site 59054, Sofia
  - Teva Investigational Site 59059, Sofia
  - Teva Investigational Site 59045, Sofia
  - Teva Investigational Site 59049, Stara Zagora
  - Teva Investigational Site 59046, Varna
  - Teva Investigational Site 59051, Veliko Tarnovo
  - Teva Investigational Site 59053, Veliko Tarnovo
- Canada (4):
  - Teva Investigational Site 11013, Edmonton, Alberta
  - Teva Investigational Site 11014, Burnaby, British Columbia
  - Teva Investigational Site 11015, Ottawa
  - Teva Investigational Site 11016, Saskatoon
- Croatia (3):
  - Teva Investigational Site 60010, Osijek
  - Teva Investigational Site 60011, Varaždin
  - Teva Investigational Site 60009, Zagreb
- Czechia (9):
  - Teva Investigational Site 54042, Brno
  - Teva Investigational Site 54043, Havířov
  - Teva Investigational Site 54047, Hradec Králové
  - Teva Investigational Site 54046, Jihlava
  - Teva Investigational Site 54044, Olomouc
  - Teva Investigational Site 54045, Ostrava
  - Teva Investigational Site 54049, Prague
  - Teva Investigational Site 54041, Prague
  - Teva Investigational Site 54048, Teplice
- Estonia (4):
  - Teva Investigational Site 55005, Pärnu
  - Teva Investigational Site 55008, Tallinn
  - Teva Investigational Site 55006, Tallinn
  - Teva Investigational Site 55007, Tartu
- France (5):
  - Teva Investigational Site 35075, Clermont-Ferrand
  - Teva Investigational Site 35077, Dijon
  - Teva Investigational Site 35073, Lille
  - Teva Investigational Site 35076, Lyon
  - Teva Investigational Site 35079, Nîmes
- Georgia (6):
  - Teva Investigational Site 81018, Tbilisi
  - Teva Investigational Site 81014, Tbilisi
  - Teva Investigational Site 81015, Tbilisi
  - Teva Investigational Site 81019, Tbilisi
  - Teva Investigational Site 81017, Tbilisi
  - Teva Investigational Site 81016, Tbilisi
- Germany (27):
  - Teva Investigational Site 32199, Bad Mergentheim
  - Teva Investigational Site 32195, Berg
  - Teva Investigational Site 32200, Berlin
  - Teva Investigational Site 32186, Berlin
  - Teva Investigational Site 32176, Berlin
  - Teva Investigational Site 32174, Berlin
  - Teva Investigational Site 32198, Berlin
  - Teva Investigational Site 32177, Bochum
  - Teva Investigational Site 32183, Cologne
  - Teva Investigational Site 32193, Dresden
  - Teva Investigational Site 32184, Erbach im Odenwald
  - Teva Investigational Site 32189, Erfurt
  - Teva Investigational Site 32203, Giessen
  - Teva Investigational Site 32202, Goettigen
  - Teva Investigational Site 32196, Halle
  - Teva Investigational Site 32181, Hamburg
  - Teva Investigational Site 32179, Hamburg
  - Teva Investigational Site 32182, Hanover
  - Teva Investigational Site 32175, Ibbenbueren
  - Teva Investigational Site 32201, Jena
  - Teva Investigational Site 32190, Leipzig
  - Teva Investigational Site 32185, Magdeburg
  - Teva Investigational Site 32191, Rostock
  - Teva Investigational Site 32194, Teupitz
  - Teva Investigational Site 32173, Ulm
  - Teva Investigational Site 32197, Wermsdorf
  - Teva Investigational Site 32188, Westerstede
- Greece (7):
  - Teva Investigational Site 63027, Athens
  - Teva Investigational Site 63024, Athens
  - Teva Investigational Site 63029, Chaïdári
  - Teva Investigational Site 63026, Heraklion
  - Teva Investigational Site 63030, Larissa
  - Teva Investigational Site 63025, Thessaloniki
  - Teva Investigational Site 63028, Thessaloniki
- Hungary (4):
  - Teva Investigational Site 51046, Budapest
  - Teva Investigational Site 51043, Debrecen
  - Teva Investigational Site 51045, Eger
  - Teva Investigational Site 51044, Kaposvár
- Israel (4):
  - Teva Investigational Site 80023, Haifa
  - Teva Investigational Site 80024, Haifa
  - Teva Investigational Site 80020, Ramat Gan
  - Teva Investigational Site 80021, Tel Aviv
- Italy (15):
  - Teva Investigational Site 30037, Bologna
  - Teva Investigational Site 30031, Castelfiorentino
  - Teva Investigational Site 30030, Cefalù
  - Teva Investigational Site 30032, Chieti
  - Teva Investigational Site 30024, Florence
  - Teva Investigational Site 30029, Gallarate
  - Teva Investigational Site 30023, Milan
  - Teva Investigational Site 30039, Milan
  - Teva Investigational Site 30034, Napoli
  - Teva Investigational Site 30027, Palermo
  - Teva Investigational Site 30028, Rome
  - Teva Investigational Site 30025, Rome
  - Teva Investigational Site 30026, Rome
  - Teva Investigational Site 30035, Rome
  - Teva Investigational Site 30040, Verona
- Latvia (2):
  - Teva Investigational Site 56006, Riga
  - Teva Investigational Site 56005, Riga
- Moldova (3):
  - Teva Investigational Site 70006, Chisinau
  - Teva Investigational Site 70005, Chisinau
  - Teva Investigational Site 70008, Chisinau
- Teva Investigational Site 66002, Podgorica, Montenegro
- North Macedonia (3):
  - Teva Investigational Site 65010, Skopje
  - Teva Investigational Site 65011, Skopje
  - Teva Investigational Site 65012, Skopje
- Poland (20):
  - Teva Investigational Site 53066, Bialystok
  - Teva Investigational Site 53071, Bialystok
  - Teva Investigational Site 53085, Bydgoszcz
  - Teva Investigational Site 53084, Częstochowa
  - Teva Investigational Site 53069, Gdansk
  - Teva Investigational Site 53083, Gdansk
  - Teva Investigational Site 53067, Gdansk
  - Teva Investigational Site 53064, Gmina Końskie
  - Teva Investigational Site 53078, Grodzisk Mazowiecki
  - Teva Investigational Site 53080, Katowice
  - Teva Investigational Site 53081, Katowice
  - Teva Investigational Site 53073, Katowice
  - Teva Investigational Site 53070, Katowice
  - Teva Investigational Site 53074, Katowice
  - Teva Investigational Site 53065, Konstancin-Jeziorna
  - Teva Investigational Site 53072, Kościerzyna
  - Teva Investigational Site 53063, Lodz
  - Teva Investigational Site 53079, Olsztyn
  - Teva Investigational Site 53068, Plewiska
  - Teva Investigational Site 53076, Szczecin
- Romania (17):
  - Teva Investigational Site 52045, Baloteşti
  - Teva Investigational Site 52041, Bucharest
  - Teva Investigational Site 52050, Bucharest
  - Teva Investigational Site 52037, Bucharest
  - Teva Investigational Site 52034, Bucharest
  - Teva Investigational Site 52040, Cluj-Napoca
  - Teva Investigational Site 52036, Cluj-Napoca
  - Teva Investigational Site 52038, Constanța
  - Teva Investigational Site 52044, Constanța
  - Teva Investigational Site 52048, Craiova
  - Teva Investigational Site 52049, Hunedoara
  - Teva Investigational Site 52042, Iași
  - Teva Investigational Site 52039, Oradea
  - Teva Investigational Site 52047, Piatra Neamţ
  - Teva Investigational Site 52046, Sibiu
  - Teva Investigational Site 52035, Târgu Mureş
  - Teva Investigational Site 52043, Timișoara
- Russia (26):
  - Teva Investigational Site 50130, Barnaul
  - Teva Investigational Site 50129, Chelyabinsk
  - Teva Investigational Site 50208, Kazan'
  - Teva Investigational Site 50148, Kemerovo
  - Teva Investigational Site 50144, Krasnodar
  - Teva Investigational Site 50147, Moscow
  - Teva Investigational Site 50124, Moscow
  - Teva Investigational Site 50133, Moscow
  - Teva Investigational Site 50146, Moscow
  - Teva Investigational Site 50141, Nizhny Novgorod
  - Teva Investigational Site 50128, Nizhny Novgorod
  - Teva Investigational Site 50131, Nizhny Novgorod
  - Teva Investigational Site 50127, Perm
  - Teva Investigational Site 50143, Rostov-on-Don
  - Teva Investigational Site 50149, Rostov-on-Don
  - Teva Investigational Site 50126, Saint Petersburg
  - Teva Investigational Site 50137, Saint Petersburg
  - Teva Investigational Site 50140, Saint Petersburg
  - Teva Investigational Site 50138, Samara
  - Teva Investigational Site 50135, Saratov
  - Teva Investigational Site 50136, Smolensk
  - Teva Investigational Site 50125, Tomsk
  - Teva Investigational Site 50139, Tyumen
  - Teva Investigational Site 50134, Ufa
  - Teva Investigational Site 50132, Volgograd
  - Teva Investigational Site 50142, Yaroslavl
- Serbia (12):
  - Teva Investigational Site 61025, Belgrade
  - Teva Investigational Site 61027, Belgrade
  - Teva Investigational Site 61024, Belgrade
  - Teva Investigational Site 61018, Čačak
  - Teva Investigational Site 61015, Kragujevac
  - Teva Investigational Site 61014, Niš
  - Teva Investigational Site 61019, Sombor
  - Teva Investigational Site 61016, Subotica
  - Teva Investigational Site 61017, Užice
  - Teva Investigational Site 61022, Valjevo
  - Teva Investigational Site 61026, Vrbas
  - Teva Investigational Site 61021, Zrenjanin
- Slovakia (2):
  - Teva Investigational Site 62012, Hlohovec
  - Teva Investigational Site 62013, Trnava
- South Korea (3):
  - Teva Investigational Site 87001, Goyang-si
  - Teva Investigational Site 87003, Seoul
  - Teva Investigational Site 87002, Seoul
- Spain (9):
  - Teva Investigational Site 31035, Barcelona
  - Teva Investigational Site 31030, Barcelona
  - Teva Investigational Site 31031, Getafe
  - Teva Investigational Site 31036, L'Hospitalet de Llobregat
  - Teva Investigational Site 31032, Madrid
  - Teva Investigational Site 31034, Madrid
  - Teva Investigational Site 31033, Navarro
  - Teva Investigational Site 31039, Oviedo
  - Teva Investigational Site 31037, Salt
- Ukraine (20):
  - Teva Investigational Site 58087, Chernihiv
  - Teva Investigational Site 58083, Chernivtsi
  - Teva Investigational Site 58077, Dnipropetrovsk
  - Teva Investigational Site 58088, Ivano-Frankivsk
  - Teva Investigational Site 58076, Ivano-Frankivsk
  - Teva Investigational Site 58116, Kharkiv
  - Teva Investigational Site 58084, Kharkiv
  - Teva Investigational Site 58089, Kiev
  - Teva Investigational Site 58073, Kyiv
  - Teva Investigational Site 58078, Kyiv
  - Teva Investigational Site 58081, Kyiv
  - Teva Investigational Site 58115, Lviv
  - Teva Investigational Site 58086, Lviv
  - Teva Investigational Site 58085, Odesa
  - Teva Investigational Site 58074, Odesa
  - Teva Investigational Site 58082, Poltava
  - Teva Investigational Site 58080, Simferopol
  - Teva Investigational Site 58072, Vinnytsia
  - Teva Investigational Site 58079, Zaporizhzhya
  - Teva Investigational Site 58075, Zaporizhzhya
- United Kingdom (7):
  - Teva Investigational Site 34015, Glasgow
  - Teva Investigational Site 34011, Liverpool
  - Teva Investigational Site 34010, Liverpool
  - Teva Investigational Site 34019, London
  - Teva Investigational Site 34016, Salford
  - Teva Investigational Site 34017, Sheffield
  - Teva Investigational Site 34013, Stoke-on-Trent

REFERENCES:
- [Derived] Comi G, Dadon Y, Sasson N, Steinerman JR, Knappertz V, Vollmer TL, Boyko A, Vermersch P, Ziemssen T, Montalban X, Lublin FD, Rocca MA, Volkinshtein R, Rubinchick S, Halevy N, Filippi M. CONCERTO: A randomized, placebo-controlled trial of oral laquinimod in relapsing-remitting multiple sclerosis. Mult Scler. 2022 Apr;28(4):608-619. doi: 10.1177/13524585211032803. Epub 2021 Aug 11. PMID 34378456

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was conducted at 215 sites in 29 countries.
Groups:
- Placebo-Controlled Phase: Placebo: Participants received 2 capsules of placebo (matched to laquinimod 0.6 milligrams [mg]) once daily orally for up to 24 months.
- Placebo-Controlled Phase: Laquinimod 0.6 mg: Participants received 1 capsule of laquinimod 0.6 mg and 1 capsule of matching placebo once daily orally for up to 24 months.
- Placebo-Controlled Phase: Laquinimod 1.2 mg: Participants received laquinimod 1.2 mg (2 capsules of laquinimod 0.6 mg each) once daily orally for up to 24 months.
- Active Treatment Phase: Laquinimod 0.6 mg: Participants who completed the placebo-controlled phase on placebo and on laquinimod 0.6 mg treatment group after 01 January 2016, received 1 capsule of laquinimod 0.6 mg and 1 capsule of matching placebo once daily orally for 24 months.
- Active Treatment Phase: Laquinimod 1.2 mg: Participants who completed the placebo-controlled phase on placebo and on laquinimod 1.2 mg treatment group prior to 01 January 2016, received laquinimod 1.2 mg (2 capsules of laquinimod 0.6 mg each) once daily orally for 24 months.
- Active Treatment Phase: Off Drug: Participants who were discontinued from treatment with laquinimod 1.2 mg during the placebo-controlled phase due to sponsor decision after 01 January 2016 continued to the active-treatment phase off drug for 24 months.
Period: Placebo-Controlled Phase (24 Months)
Arm/Group | Placebo-Controlled Phase: Placebo | Placebo-Controlled Phase: Laquinimod 0.6 mg | Placebo-Controlled Phase: Laquinimod 1.2 mg | Active Treatment Phase: Laquinimod 0.6 mg | Active Treatment Phase: Laquinimod 1.2 mg | Active Treatment Phase: Off Drug
Started | 740 | 727 | 732 | 0 | 0 | 0
Completed | 596 | 623 | 532 | 0 | 0 | 0
Not Completed | 144 | 104 | 200 | 0 | 0 | 0
Not completed — Adverse Event | 8 | 13 | 9 | 0 | 0 | 0
Not completed — Lack of Efficacy | 10 | 3 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 88 | 68 | 154 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Pregnancy | 12 | 5 | 9 | 0 | 0 | 0
Not completed — Lost to Follow-up | 10 | 4 | 9 | 0 | 0 | 0
Not completed — Death | 2 | 1 | 1 | 0 | 0 | 0
Not completed — Noncompliance with drug administration | 2 | 1 | 6 | 0 | 0 | 0
Not completed — Other than specified | 11 | 9 | 10 | 0 | 0 | 0
Period: Active Treatment Phase (24 Months)
Arm/Group | Placebo-Controlled Phase: Placebo | Placebo-Controlled Phase: Laquinimod 0.6 mg | Placebo-Controlled Phase: Laquinimod 1.2 mg | Active Treatment Phase: Laquinimod 0.6 mg | Active Treatment Phase: Laquinimod 1.2 mg | Active Treatment Phase: Off Drug
Started | 0 | 0 | 0 | 891 | 504 | 215
Completed | 0 | 0 | 0 | 7 | 10 | 0
Not Completed | 0 | 0 | 0 | 884 | 494 | 215
Not completed — Adverse Event | 0 | 0 | 0 | 4 | 1 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 3 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 58 | 220 | 32
Not completed — Pregnancy | 0 | 0 | 0 | 2 | 5 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 5 | 11 | 1
Not completed — Death | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Other than specified | 0 | 0 | 0 | 1 | 5 | 2
Not completed — Noncompliance | 0 | 0 | 0 | 0 | 4 | 2
Not completed — Study terminated by sponsor | 0 | 0 | 0 | 809 | 243 | 174
Not completed — Participant withdrew per Sponsor request | 0 | 0 | 0 | 0 | 4 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) analysis set included all randomized participants.
Groups:
- Placebo-Controlled Phase: Placebo: Participants received 2 capsules of placebo (matched to laquinimod 0.6 mg) once daily orally for up to 24 months.
- Total: Total of all reporting groups
Arm/Group | Placebo-Controlled Phase: Placebo | Placebo-Controlled Phase: Laquinimod 0.6 mg | Placebo-Controlled Phase: Laquinimod 1.2 mg | Total
Number analyzed (Participants) | 740 | 727 | 732 | 2199
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.9 (8.95) | 36.8 (9.25) | 36.1 (9.22) | 36.3 (9.14)
Age, Customized [Count of Participants; unit: Participants]
  Adults (18-64 years) | 740 | 727 | 732 | 2199
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 488 | 510 | 475 | 1473
  Male | 252 | 217 | 257 | 726
Race [Count of Participants; unit: Participants]
  White | 724 | 712 | 717 | 2153
  Black | 3 | 3 | 3 | 9
  Asian | 3 | 2 | 3 | 8
  Other | 10 | 8 | 9 | 27
  Missing | 0 | 2 | 0 | 2
Kurtzke's Expanded Disability Status Scale (EDSS) Score [Count of Participants; unit: Participants] — EDSS assesses disability in 8 functional systems with an overall score ranging from 0 (normal) to 10 (death due to multiple sclerosis [MS]).
  Participants
    Less than or equal to (<=) 4.0 | 653 | 635 | 644 | 1932
    Greater than (>) 4.0 | 87 | 90 | 88 | 265
    Missing | 0 | 2 | 0 | 2
Normalized Brain Volume [Mean (Standard Deviation); unit: milliliters (mL)] — Population: This characteristic was analyzed for a total of 2187 participants (Placebo [737], Laquinimod 0.6 mg [722], and Laquinimod 1.2 mg [728])
  milliliters (mL)
    number analyzed (Participants) | 737 | 722 | 728 | 2187
    (all) | 1437.2 (93.37) | 1433.0 (92.49) | 1434.4 (93.41) | 1434.9 (93.07)

OUTCOME MEASURES:

1. Primary Outcome: Placebo-Controlled Phase: Time to Confirmed Disease Progression (CDP) Confirmed After At Least 3 Months (Number of Participants With CDP After At Least 3 Months)
Description: Time to CDP was defined as the time to a sustained increase in Kurtzke's Expanded Disability Status Scale (EDSS) score of at least 1 point if baseline EDSS score was less than or equal to 5.0, or at least 0.5 point if the baseline EDSS score was 5.5, over a period of at least three months. EDSS assesses disability in 8 functional systems with an overall score ranging from 0 (normal) to 10 (death due to multiple sclerosis [MS]). Data is presented as distribution of CDP (number of participants with CDP) sustained for 3 months.
Time Frame: Baseline to Month 24
Population: ITT analysis set included all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo-Controlled Phase: Placebo | Placebo-Controlled Phase: Laquinimod 0.6 mg | Placebo-Controlled Phase: Laquinimod 1.2 mg
Number analyzed (Participants) | 740 | 727 | 732
Participants | 73 | 66 | 69
Statistical Analysis 1: Comparison: Placebo-Controlled Phase: Placebo vs Placebo-Controlled Phase: Laquinimod 0.6 mg; The primary analysis for the comparison between laquinimod 0.6 mg versus placebo was conducted using the baseline adjusted Cox proportional hazards model. Categorical EDSS at baseline (less than or equal to [<=] 4 or greater than [>] 4), country/geographical region (CGR), categorical age at baseline (<=38 or >38), and T2 volume at baseline were included as covariates in the model; Test type: Superiority; p = 0.7057, Cox proportional hazards model — Threshold for significance at 0.05 level; Hazard Ratio (HR) = 0.937, 95% CI 2-sided [0.668 to 1.313]

2. Secondary Outcome: Placebo-Controlled Phase: Percent Change From Baseline in Brain Volume at Month 15
Description: Brain atrophy was defined by the percent change in brain volume from baseline to Month 15. For participants who prematurely discontinued treatment or completed the placebo-controlled phase before Month 15, the last available measurement was used, provided it was performed at least 9 months following the initiation of study drug.
Time Frame: Baseline, Month 15
Population: The modified intent-to-treat 1 (mITT1) analysis set included data from all randomized participants at the Month 15 visit. Here, 'Overall number of participants analyzed' = Participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo-Controlled Phase: Placebo | Placebo-Controlled Phase: Laquinimod 0.6 mg | Placebo-Controlled Phase: Laquinimod 1.2 mg
Number analyzed (Participants) | 619 | 636 | 616
percent change | -0.8 (1.02) [lower limit 1.02] | -0.4 (1.01) [lower limit 1.01] | -0.4 (1.05) [lower limit 1.05]

3. Secondary Outcome: Placebo-Controlled Phase: Time to First Confirmed Relapse (Number of Participants With Confirmed Relapse)
Description: Relapse was defined as appearance of one or more new neurological abnormalities or reappearance or worsening of one or more previously observed neurological abnormalities, lasting for at least 48 hours (in absence of fever or any infection) and immediately preceded by an improving neurological state of at least 30 days from onset of previous relapse. An event was counted as a relapse only when the participant's symptoms were accompanied by observed objective neurological changes, consistent with an increase of at least 0.5 in EDSS; or one grade in score of 2 or more of 7 Functional Systems (FS) (excluding changes in bowel or bladder function or cognition); or 2 grades in score of one of the FS as compared to previous evaluation. EDSS assesses disability in 8 FS with an overall score ranging from 0 (normal) to 10 (death due to MS). Data is presented as distribution of relapsing participants (number of participants with confirmed relapse).
Time Frame: Baseline to Month 24
Population: ITT analysis set included all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo-Controlled Phase: Placebo | Placebo-Controlled Phase: Laquinimod 0.6 mg | Placebo-Controlled Phase: Laquinimod 1.2 mg
Number analyzed (Participants) | 740 | 727 | 732
Participants | 332 | 269 | 222

4. Secondary Outcome: Placebo-Controlled Phase: Time to CDP Confirmed After At Least 6 Months (Number of Participants With CDP After At Least 6 Months)
Description: Time to CDP was defined as the time to a sustained increase in Kurtzke's EDSS score of at least 1 point if baseline EDSS score was less than or equal to 5.0, or at least 0.5 point if the baseline EDSS score was 5.5, over a period of at least 6 months. EDSS assesses disability in 8 functional systems with an overall score ranging from 0 (normal) to 10 (death due to MS). Data is presented as distribution of CDP (number of participants with CDP) sustained for 6 months.
Time Frame: Baseline to Month 24
Population: ITT analysis set included all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo-Controlled Phase: Placebo | Placebo-Controlled Phase: Laquinimod 0.6 mg | Placebo-Controlled Phase: Laquinimod 1.2 mg
Number analyzed (Participants) | 740 | 727 | 732
Participants | 49 | 49 | 51

5. Secondary Outcome: Placebo-Controlled Phase: Time to CDP Confirmed After At Least 9 Months (Number of Participants With Confirmed Relapse After At Least 9 Months)
Description: Time to CDP was defined as the time to a sustained increase in Kurtzke's EDSS score of at least 1 point if baseline EDSS score was less than or equal to 5.0, or at least 0.5 point if the baseline EDSS score was 5.5, over a period of at least 9 months. EDSS assesses disability in 8 functional systems with an overall score ranging from 0 (normal) to 10 (death due to MS). Data is presented as distribution of CDP (number of participants with CDP) sustained for 9 months.
Time Frame: Baseline to Month 24
Population: ITT analysis set included all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo-Controlled Phase: Placebo | Placebo-Controlled Phase: Laquinimod 0.6 mg | Placebo-Controlled Phase: Laquinimod 1.2 mg
Number analyzed (Participants) | 740 | 727 | 732
Participants | 38 | 38 | 39

6. Other Pre Specified Outcome: Placebo-Controlled Phase: Number of Participants With Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. AEs included both SAEs and non-serious AEs.
Time Frame: Baseline up to Month 24
Population: Safety analysis set included all participants who were randomized and received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo-Controlled Phase: Placebo | Placebo-Controlled Phase: Laquinimod 0.6 mg | Placebo-Controlled Phase: Laquinimod 1.2 mg
Number analyzed (Participants) | 740 | 727 | 732
Participants | 546 | 565 | 575

7. Other Pre Specified Outcome: Active-Treatment Phase: Number of Participants With AEs
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. AEs included both SAEs and non-serious AEs.
Time Frame: Baseline (Month 0 of active-treatment phase/Month 24 of placebo-controlled phase) up to Month 24 of active-treatment phase
Population: Safety analysis set in active-treatment phase included all participants who completed placebo-controlled phase on treatment and continued to either of the 2 laquinimod treatments during active-treatment phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Active Treatment Phase: Laquinimod 0.6 mg | Active Treatment Phase: Laquinimod 1.2 mg
Number analyzed (Participants) | 891 | 504
Participants | 442 | 241

8. Other Pre Specified Outcome: Placebo-Controlled Phase: Number of Participants With Clinically Significant Vital Signs Abnormalities
Description: Clinically significant vital signs abnormalities included: Pulse rate: greater than or equal to (>=) 120 beats per minute (bpm) and increase from baseline of >=30 bpm, <=45 bpm and decrease from baseline of >=30 bpm; Systolic blood pressure: >=180 millimeters of mercury (mmHg) and increase from baseline of >=30 mmHg, <=90 and decrease from baseline of >=30 mmHg; Diastolic blood pressure: >=100 mmHg and increase from baseline of >=20 mmHg, <=50 mmHg and decrease from baseline of >=20 mmHg.
Time Frame: Baseline up to Week 24
Population: Safety analysis set included all participants who were randomized and received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo-Controlled Phase: Placebo | Placebo-Controlled Phase: Laquinimod 0.6 mg | Placebo-Controlled Phase: Laquinimod 1.2 mg
Number analyzed (Participants) | 740 | 727 | 732
Participants | 21 | 21 | 29

9. Other Pre Specified Outcome: Active-Treatment Phase: Number of Participants With Clinically Significant Vital Signs Abnormalities
Description: Clinically significant vital signs abnormalities included: Pulse rate: >=120 bpm and increase from baseline of >=30 bpm, <=45 bpm and decrease from baseline of >=30 bpm; Systolic blood pressure: >=180 mmHg and increase from baseline of >=30 mmHg, <=90 and decrease from baseline of >=30 mmHg; Diastolic blood pressure: >=100 mmHg and increase from baseline of >=20 mmHg, <=50 mmHg and decrease from baseline of >=20 mmHg.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Active Treatment Phase: Laquinimod 0.6 mg | Active Treatment Phase: Laquinimod 1.2 mg
Number analyzed (Participants) | 891 | 504
Participants | 17 | 7

10. Other Pre Specified Outcome: Placebo-Controlled Phase: Number of Participants With Shift From Baseline to Endpoint in Electrocardiogram (ECG) Parameters
Description: ECG parameters included: PR interval, QRS interval, QT interval corrected using the Fridericia formula (QTcF) and QT interval corrected using the Bazett's formula (QTcB). Shifts represented as Baseline - endpoint value (last observed post-baseline value). Abnormal NCS indicated an abnormal but not clinically significant finding. Abnormal CS indicated an abnormal and clinically significant finding.
Time Frame: Baseline, Endpoint (Month 24)
Population: Safety analysis set included all participants who were randomized and received at least one dose of study drug. Here, 'Overall number of participants analyzed=participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo-Controlled Phase: Placebo | Placebo-Controlled Phase: Laquinimod 0.6 mg | Placebo-Controlled Phase: Laquinimod 1.2 mg
Number analyzed (Participants) | 734 | 723 | 724
Participants
  Normal - Normal | 463 | 467 | 470
  Normal - Abnormal NCS | 139 | 124 | 126
  Normal - Abnormal CS | 0 | 6 | 5
  Abnormal NCS - Normal | 32 | 27 | 28
  Abnormal NCS - Abnormal NCS | 98 | 96 | 90
  Abnormal NCS - Abnormal CS | 1 | 1 | 2
  Abnormal CS - Normal | 0 | 1 | 0
  Abnormal CS - Abnormal NCS | 0 | 0 | 0
  Abnormal CS - Abnormal CS | 1 | 1 | 3

11. Other Pre Specified Outcome: Active Treatment Phase: Number of Participants With Shift From Baseline to Endpoint in ECG Parameters
Description: ECG parameters included: PR interval, QRS interval, QTcF and QTcB. Shifts represented as Baseline - endpoint value (last observed post-baseline value). Abnormal NCS indicated an abnormal but not clinically significant finding. Abnormal CS indicated an abnormal and clinically significant finding.
Time Frame: Baseline (Month 0 of active-treatment phase/Month 24 of placebo-controlled phase), endpoint (Month 24 of active-treatment phase)
Population: Safety analysis set in active-treatment phase included all participants who completed placebo-controlled phase on treatment and continued to either of the 2 laquinimod treatments during active-treatment phase and had ECG shift from baseline data available.
Measure: Count of Participants; unit: Participants
Arm/Group | Active Treatment Phase: Laquinimod 0.6 mg | Active Treatment Phase: Laquinimod 1.2 mg
Number analyzed (Participants) | 888 | 501
Participants
  Normal - Normal | 641 | 353
  Normal - Abnormal NCS | 137 | 80
  Normal - Abnormal CS | 7 | 5
  Abnormal NCS - Normal | 18 | 17
  Abnormal NCS - Abnormal NCS | 81 | 45
  Abnormal NCS - Abnormal CS | 4 | 0
  Abnormal CS - Normal | 0 | 0
  Abnormal CS - Abnormal NCS | 0 | 0
  Abnormal CS - Abnormal CS | 0 | 1

12. Other Pre Specified Outcome: Placebo-Controlled Phase: Number of Participants With Potentially Clinically Significant Abnormal Serum Chemistry
Description: Potentially clinically significant serum chemistry abnormalities included: Glucose <=3 and >=13.88 millimoles per liter (mmol/L); Alanine aminotransferase (ALT) (in units per liter [U/L]), aspartate aminotransferase (AST) (in U/L), alkaline phosphatase (in U/L), gamma-glutamyltransferase (GGT) (in U/L), creatine phosphokinase (CPK) (in U/L), C-reactive protein (CRP) (in milligrams per liter [mg/L]), pancreatic amylase (in U/L)>=3 * upper limit of normal (ULN); Fibrinogen >=6 grams per liter (gm/L); Sodium <=130 and >=150 mmol/L; Potassium <=3.2 and >=5.5 mmol/L; Calcium <=1.87 and >=2.75 mmol/L; Phosphate <=0.65 and >=1.61 mmol/L.
Time Frame: Baseline up to Month 24
Population: Safety analysis set included all participants who were randomized and received at least one dose of study drug. Here, 'Overall number of participants analyzed'=participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo-Controlled Phase: Placebo | Placebo-Controlled Phase: Laquinimod 0.6 mg | Placebo-Controlled Phase: Laquinimod 1.2 mg
Number analyzed (Participants) | 736 | 723 | 724
Participants | 157 | 165 | 187

13. Other Pre Specified Outcome: Active Treatment Phase: Number of Participants With Potentially Clinically Significant Abnormal Serum Chemistry
Description: Potentially clinically significant serum chemistry abnormalities included: Glucose <=3 and >=13.88 mmol/L; ALT (in U/L), AST (in U/L), alkaline phosphatase (in U/L), GGT (in U/L), CPK (in U/L), CRP (in mg/L), pancreatic amylase (in U/L)>=3 * ULN; Fibrinogen >=6 gm/L; Sodium <=130 and >=150 mmol/L; Potassium <=3.2 and >=5.5 mmol/L; Calcium <=1.87 and >=2.75 mmol/L; Phosphate <=0.65 and >=1.61 mmol/L; Blood urea nitrogen (in mmol/L); Total bilirubin >=28 micromols per liter (micromols/L); Creatinine >=117 micromols/L; Albumin <=25 gm/L.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Active Treatment Phase: Laquinimod 0.6 mg | Active Treatment Phase: Laquinimod 1.2 mg
Number analyzed (Participants) | 891 | 504
Participants | 887 | 501

14. Other Pre Specified Outcome: Placebo-Controlled Phase: Number of Participants With Potentially Clinically Significant Abnormal Hematology Values
Description: Potentially clinically significant hematological abnormalities included: Hemoglobin <=11.5 grams per deciliter (gm/dL) in males and <=10 gm/dL in females; White blood cells (WBCs) count <=2.5 and >=21*10^9 per liter (L); Absolute neutrophil count (ANC) <=1.49*10^9 per L; Platelet count <=100 and >=600*10^9 per L.
Time Frame: Baseline up to Month 24
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo-Controlled Phase: Placebo | Placebo-Controlled Phase: Laquinimod 0.6 mg | Placebo-Controlled Phase: Laquinimod 1.2 mg
Number analyzed (Participants) | 735 | 723 | 723
Participants | 71 | 78 | 83

15. Other Pre Specified Outcome: Active Treatment Phase: Number of Participants With Potentially Clinically Significant Abnormal Hematology Values
Description: Potentially clinically significant hematological abnormalities included: Hemoglobin <=11.5, >=20 gm/dL in males, and <=10, >=18.5 gm/dL in females; WBCs count <=2.5 and >=21*10^9 per L; ANC <=1.49*10^9 per L; Platelet count <=100 and >=600*10^9 per L.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Active Treatment Phase: Laquinimod 0.6 mg | Active Treatment Phase: Laquinimod 1.2 mg
Number analyzed (Participants) | 891 | 504
Participants | 886 | 499

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the procedure and at each follow-up visit at 2 weeks, 6 weeks, 12 weeks, 24 weeks, and 52 weeks post-treatment.
Groups:
- Active Treatment Phase: Early Laquinimod 0.6 mg: Participants who completed the placebo-controlled phase on laquinimod 0.6 mg treatment group after 01 January 2016, received 1 capsule of laquinimod 0.6 mg and 1 capsule of matching placebo once daily orally for 24 months.
- Active Treatment Phase: Early Laquinimod 1.2 mg: Participants who completed the placebo-controlled phase on laquinimod 1.2 mg treatment group prior to 01 January 2016, received laquinimod 1.2 mg (2 capsules of laquinimod 0.6 mg each) once daily orally for 24 months.
- Active Treatment Phase: Off Drug: Participants who were discontinued from treatment with laquinimod 1.2 mg during the placebo-controlled phase due to sponsor decision after 01 January 2016, continued to the active-treatment phase off drug for 24 months.
- Active Treatment Phase: From Placebo to Laquinimod 0.6 mg: Participants who completed the placebo-controlled phase on placebo treatment group after 01 January 2016, received 1 capsule of laquinimod 0.6 mg and 1 capsule of matching placebo once daily orally for 24 months.
- Active Treatment Phase: From Placebo to Laquinimod 1.2 mg: Participants who completed the placebo-controlled phase on placebo treatment group prior to 01 January 2016, received laquinimod 1.2 mg (2 capsules of laquinimod 0.6 mg each) once daily orally for 24 months.
Arm/Group | Placebo-Controlled Phase: Laquinimod 0.6 mg | Placebo-Controlled Phase: Laquinimod 1.2 mg | Placebo-Controlled Phase: Placebo | Active Treatment Phase: Early Laquinimod 0.6 mg | Active Treatment Phase: Early Laquinimod 1.2 mg | Active Treatment Phase: Off Drug | Active Treatment Phase: From Placebo to Laquinimod 0.6 mg | Active Treatment Phase: From Placebo to Laquinimod 1.2 mg
All-Cause Mortality (participants affected / at risk) | 1/727 | 1/732 | 2/740 | 2/580 | 0/268 | 0/215 | 0/311 | 0/236
Serious Adverse Events (participants affected / at risk) | 57/727 | 49/732 | 43/740 | 24/580 | 10/268 | 5/215 | 5/311 | 9/236
Other Adverse Events (participants affected / at risk) | 262/727 | 286/732 | 243/740 | 102/580 | 46/268 | 35/215 | 43/311 | 43/236
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo-Controlled Phase: Laquinimod 0.6 mg (N=727) | Placebo-Controlled Phase: Laquinimod 1.2 mg (N=732) | Placebo-Controlled Phase: Placebo (N=740) | Active Treatment Phase: Early Laquinimod 0.6 mg (N=580) | Active Treatment Phase: Early Laquinimod 1.2 mg (N=268) | Active Treatment Phase: Off Drug (N=215) | Active Treatment Phase: From Placebo to Laquinimod 0.6 mg (N=311) | Active Treatment Phase: From Placebo to Laquinimod 1.2 mg (N=236)
Hypochromic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiovascular insufficiency (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coeliac disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Duodenal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric polyps (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatic necrosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis chronic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periodontal inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritoneal adhesions (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Strangulated hernia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis chronic (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis obstructive (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis cholestatic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sarcoidosis (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess oral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis infective (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endometritis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterovirus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Helicobacter gastritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis B (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster oticus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infected dermal cyst (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ovarian abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pilonidal cyst (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis chronic (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Salpingitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Salpingo-oophoritis (Infections and infestations) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary bladder abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bone contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brain contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cartilage injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jaw fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Poisoning deliberate (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postoperative adhesion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pubis fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skull fractured base (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Traumatic liver injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alpha 1 foetoprotein abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nuclear magnetic resonance imaging brain abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metabolic disorder (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femoroacetabular impingement (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign neoplasm of adrenal gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metastases to chest wall (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Salivary gland adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coma (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple sclerosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple sclerosis relapse (Nervous system disorders) | 2 (2) | 1 (1) | 7 (7) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neurological decompensation (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuromyelitis optica spectrum disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psychomotor hyperactivity (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Trigeminal neuralgia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foetal growth abnormality (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Unintended pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute psychosis (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Affective disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Major depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Persecutory delusion (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Personality change due to a general medical condition (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Schizophrenia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acquired hydrocele (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adnexal torsion (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervix disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fallopian tube cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Menometrorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ovarian haemorrhage (Reproductive system and breast disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Polycystic ovaries (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vasomotor rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hospitalisation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Embolism arterial (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Varicose vein (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vasculitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Autoimmune pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis toxic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tuberculosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intentional overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Status epilepticus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abortion (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abortion threatened (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Completed suicide (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo-Controlled Phase: Laquinimod 0.6 mg (N=727) | Placebo-Controlled Phase: Laquinimod 1.2 mg (N=732) | Placebo-Controlled Phase: Placebo (N=740) | Active Treatment Phase: Early Laquinimod 0.6 mg (N=580) | Active Treatment Phase: Early Laquinimod 1.2 mg (N=268) | Active Treatment Phase: Off Drug (N=215) | Active Treatment Phase: From Placebo to Laquinimod 0.6 mg (N=311) | Active Treatment Phase: From Placebo to Laquinimod 1.2 mg (N=236)
Anaemia (Blood and lymphatic system disorders) | 28 (32) | 43 (50) | 30 (35) | 22 (25) | 13 (16) | 7 (7) | 9 (9) | 9 (12)
Nasopharyngitis (Infections and infestations) | 63 (90) | 60 (86) | 63 (91) | 40 (52) | 14 (20) | 8 (13) | 11 (13) | 11 (13)
Respiratory tract infection viral (Infections and infestations) | 32 (54) | 31 (37) | 39 (56) | 14 (19) | 7 (9) | 3 (3) | 3 (3) | 5 (6)
Amylase increased (Investigations) | 17 (20) | 38 (43) | 18 (19) | 6 (7) | 2 (2) | 2 (2) | 6 (6) | 5 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 54 (74) | 85 (110) | 39 (47) | 12 (14) | 8 (10) | 9 (10) | 1 (1) | 12 (14)
Headache (Nervous system disorders) | 122 (238) | 131 (227) | 116 (222) | 22 (38) | 8 (14) | 10 (13) | 14 (25) | 10 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.